CLINICAL TRIAL: NCT03318601
Title: Evaluation of Copeptin in Patients With Cirrhosis and Ascites
Acronym: CIRCOPEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIRCOPEP study
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Cirrhotic Patients With Ascites
Keywords: cirrhotic; ascite; copeptin
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: cirrhotic patients with ascites requiring prolonged hospitalization in the Hepato-gastroenterology departments of the Besançon, Nancy and Reims hospitals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cirrhotic patients with ascites (Experimental): cirrhotic patients with ascites requiring prolonged hospitalization
  Interventions: Procedure: Blood taking

INTERVENTIONS:
Procedure: Blood taking — Blood taking in 2 times :
  * J0 : 15 mL
  * J14 : 5 mL 20 mL in total volume

SUMMARY:
Copeptin is a glycopeptide released by the post-pituitary gland. In case of decrease in blood volume or blood pressure, it is secreted in the serum in an equimolar quantity to arginine vasopressin (AVP) . Unlike AVP, copeptin is readily assayable in serum and its prognostic value has been recently observed during cirrhosis. However, the pathophysiological relationships between serum copeptin concentrations and indirect markers of inflammation are unknown.

The main objective of this multicenter pilot study is to study the relationship between serum copeptin and markers of inflammatory stress in cirrhotic patients with ascites. It is indeed in this population with high-risk of complications that most need biomarkers of events (like death) are needed. The main secondary objective is to evaluate the prognostic interest at 6 months of the variation of copeptin between day 0- day15.

DETAILED DESCRIPTION:
The investigators wish to include prospectively 100 cirrhotic patients with ascites requiring prolonged hospitalization in the Hepato-gastroenterology departments of the Besançon, Nancy and Reims hospitals. The inclusion and follow-up periods will be six months each. At the inclusion of the patients we will evaluate the correlations between the plasma concentration of copeptin and 1 / the severity of cirrhosis (Child-Pugh and MELD scores) and serum sodium; 2 / systemic inflammation markers (CRP, leukocytes, IL-6 and lipopolysaccharides), 3 / calprotectin concentration in ascites. "

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Age between 18 and 80 years
* Acute decompensation of cirrhosis with occurrence of ascites
* Hospitalisationfor a complication of cirrhosis (first occurrence of ascites or recurrent ascites requiring hospitalization, gastrointestinal bleeding, hepatic encephalopathy, etc..)
* Patients participating to Ca-DRISLA study
* Information and Consent form signed

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Age minor to 18 years
* Age major to 80 years
* Adult under protection law
* outpatients hospitalized for paracentesis
* ascites not related to portal hypertension (pancreatic ascites, peritoneal carcinosis…) Patients with hepatocellular carcinoma could be included

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05-09 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Correlation between copetine and other biomarkers | Day 0
  Correlation will be studied with the Spearmann or Pearson' correlation coefficient
Correlation between copetine and other biomarkers | Day 7
  Correlation will be studied with the Spearmann or Pearson' correlation coefficient
Correlation between copetine and other biomarkers | Day 15
  Correlation will be studied with the Spearmann or Pearson' correlation coefficient

SECONDARY OUTCOMES:
Performance of CRP | Day 0
  ROC curve
Performance of IL-6 | Day 0
  ROC curve
Performance of LPS | Day 0
  ROC curve
Performance of copeptine | Day 0
  ROC curve
Copetine variation | Day 15
  pronostic interest
Copetine concentrations | Day 0
  Compared betwenn cirhotic patient and healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No